CLINICAL TRIAL: NCT06132698
Title: Efficacy and Safety of Immune Checkpoint (PD-1) Inhibitor Combined With Pemetrexed Intrathecal Injection in Patients With Leptomeningeal Metastases in NSCLC
Brief Title: Immune Checkpoint Inhibitors Intrathecal Injection in Patients With Leptomeningeal Metastases in NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ting Liu, Clinical Investigator, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: West China Hospital of SU
Record Dates: First submitted 2023-11-07; First posted 2023-11-15 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: NSCLC Associated With Leptomeningeal Metastases
MeSH Terms: interventions — tislelizumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enrolled patients were treated with an immune checkpoint inhibitor combined with pemetrexed intrathe (Experimental)
  Interventions: Drug: Tislelizumab, pemetrexed

INTERVENTIONS:
Drug: Tislelizumab, pemetrexed — Drug 1: Tislelizumab 50 mg; Drug 2: pemetrexed 20mg. intrathecal injection therapy

SUMMARY:
This is a prospective, single-arm, open clinical study, which was designed to evaluate the efficacy and safety of an immune checkpoint inhibitor combined with pemetrexed intrathecal injection in the treatment of patients with NSCLC associated with leptomeningeal metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old, male or female;
2. Patients with pathologically diagnosed non-small cell lung cancer with cerebrospinal fluid and/or MRI diagnosis of leptomeningeal metastasis;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2;
4. Expected survival time of at least 4 weeks;
5. Oncologist clarification of the potential necessity of receiving systemic therapy for metastatic tumors outside the CNS;
6. Previous radiation therapy, including whole brain radiation, stereotactic radiosurgery, or stereotactic body radiation therapy (SBRT), which must be completed at least 7 days prior to the start of treatment;
7. Patients who have received approved targeted therapies (EGFR inhibitors, ALK inhibitors, or other targeted therapeutic agents), and other systemic therapies will be allowed to remain on concurrent therapy; concurrent intrathecal therapy with other agents will not be allowed.
8. Laboratory test indicators meet the following criteria:

   1. Bone marrow function: hemoglobin (Hb) ≥80g/L; white blood cell count (WBC) ≥lower limit of normal; absolute neutrophil count (ANC) ≥1.5×10^9 /L; platelet count ≥70×109 /L;
   2. Renal function: Cr ≤ ULN (upper limit of normal) × 1.5, endogenous creatinine clearance (Ccr) ≥ 55 ml/min;
   3. Liver function: total bilirubin ≤ ULN × 1.5; ALT and AST ≤ ULN × 2.5; (if there is liver metastasis, total bilirubin is not higher than 3 times the upper limit of normal, and transaminases are not higher than 5 times the upper limit of normal);
   4. Coagulation function: international normalized ratio of prothrombin time ≤ ULN × 1.5, and partial thromboplastin time within the normal value;
9. Females of child-bearing potential agree to use contraception during the study period and for 6 months after the completion of the study; patients who have had a negative serum or urine pregnancy test within seven days prior to enrollment in the study and who are not breastfeeding; and males agreeing to use contraception during the study period and for 6 months after the completion of the study;
10. Those who have not participated in another drug clinical trial within 4 weeks prior to enrollment;
11. Subjects who can understand the study situation and voluntarily sign the informed consent form;
12. Patients are expected to be compliant and able to follow up on efficacy and adverse events according to protocol requirements.

Exclusion Criteria:

1. Diagnosis of other malignant tumors (except carcinoma in situ, basal cell carcinoma, etc.) within the previous 5 years;
2. History of allergy to pemetrexed and ICIs therapy;
3. Any previous intrathecal injection therapy;
4. Rule out differential diagnosis of LM:a. Aseptic meningitis b. Viral meningitis c. Bacterial meningitis;
5. Participation in other clinical trials or observation periods;
6. Clinical conditions that would interfere with the evaluation or interpretation of safety or findings, or impede the understanding of informed consent and compliance with protocol requirements;
7. Presence of any treatment-related toxicity from prior systemic antitumor therapy other than alopecia that does not meet CTCAE grade 1 (based on CTCAE 5.0);
8. Presence of any active autoimmune disease or history of autoimmune disease; immunodeficiency, active tuberculosis, hepatitis B ( hepatitis B virus titer HBV-DNA <500 IU/ml after treatment and if liver function is normal will be allowed), or positive test for hepatitis C virus.
9. Either disease resulting in permanent immunosuppression or requiring permanent immunosuppressive therapy;
10. Presence of active infection or serious comorbidities;
11. uncontrolled epilepsy, neurologic failure, or severe neurologic impairment related to treatment;
12. Presence of hereditary or acquired bleeding and thrombotic tendencies;
13. History of severe injury or surgery within 1 month prior to enrollment;
14. Treatment with a live or attenuated vaccine used for the prevention of infectious diseases within 30 days prior to the first administration (injectable seasonal influenza vaccine is permitted);
15. Inability to complete an enhanced MRI;
16. Treatment with immunosuppressive drugs or corticosteroids (> 10 mg prednisone or equivalent per day) within 14 days prior to enrollment; patients are allowed to receive steroid therapy to control CNS-related symptoms, but the dose must ≤ 5 mg per day of dexamethasone (or equivalent); in the absence of an active autoimmune disease, inhaled or topical steroids and adrenal gland replacement dosing are acceptable; alternative therapies (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) are permitted; patients with experimental medications that require premedication with corticosteroids are not restricted;
17. Individuals considered by the investigator to be unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (LM ORR) for leptomeningeal metastases. | 12 months.
  Defined as the response to treatment as assessed by the investigator based on the modified Response Assessment in Neuro-Oncology Leptomeningeal Metastases (RANO-LM) criteria, containing cases of complete response, partial response, and major response.

SECONDARY OUTCOMES:
Median Progression-Free Survival (CNS-PFS) in the Central Nervous System. | Time from the start of intrathecal therapy to radiologic, cytologic, or LM-related clinical progression, whichever outcome occurs first, assessed up to 12 months.
  Progression-free survival will be measured as time to radiologic, cytologic, or LM-related clinical progression.
Progression-Free Survival (PFS). | Time from the first day of administration of study drug until the first efficacy assessment of disease progression (PD) or death from any cause, assessed up to 12 months.
  Progression-free survival will be measured as time to either progression or death.
Overall survival (OS). | Time from the date of randomisation to the date of death from any cause, assessed up to 12 months.
  Overall survival will be measured as time to death from any cause.
Disease Control Rate (DCR). | 12 months.
  The DCR was defined as the proportion of patients with the best efficacy (complete response or partial response or stable disease).
Adverse events. | 12 months.
  toxicity values caused by intrathecal injection treatment.